CLINICAL TRIAL: NCT06038266
Title: Predictors of Hospital Readmission for Patients Undergoing Cardiac Surgeries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Fathy Abdelhafeez Soliman, Mr., Assiut University
Other Study IDs: PHR for Cardiac Surgery
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Surgery, Readmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac surgeries — predict perioperative risk factors for readmission after cardiac surgeries

SUMMARY:
This study aimed to identify the predictors of hospital readmission for patients undergoing cardiac surgeries.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are conditions of the heart and blood vessels that lead to significant morbidity and mortality, burden the global public health system, and are the main cause of death worldwide. CVD accounted for approximately 19.05 million global deaths in 2020. CVD is listed as the first underlying cause of death, with more than 800000 deaths in the United States in 2019. Between 2015 and 2018, 126.9 million US adults had some form of CVD. Between 2017 and 2018, direct and indirect costs of total CVD were $378.0 billion ($226.2. billion in direct costs and $151.8 billion in lost productivity/mortality).

Cardiac surgery continues to play an important role in the management of various cardiovascular disorders, including the treatment of seriously and critically ill patients. The most frequently performed procedures include coronary artery bypass graft (CABG) and valvular surgery. According to the Society of Thoracic Surgeons, the number of cardiac surgeries exceeds 300000 procedures in 2019 in the United States. Despite tremendous advancements in cardiac surgery over the past few years, postoperative hospital readmissions after cardiac surgeries still present significant challenges.

Readmission occurs when a patient is admitted to the same or a different hospital after being discharged from the relevant hospital and placed in a non-acute setting, such as his home, within a predetermined amount of time. Readmission within 30 days of adult cardiac surgery is a difﬁcult and costly problem, with rates ranging from 8% to 21%. In addition to delayed return to activities of daily living and reduced quality of life, readmission is associated with a ﬁnancial cost for patients and healthcare facilities. Increased facility costs can be substantial, especially when combined with reimbursement penalties, the cost of skilled care, and potential legal expenses.

Readmission after cardiac surgery is common and moderately predictable. According to a study done in a multi-institutional hospital in Ontario, Canada on patients who underwent CABG and/or valve surgery from 2008 to 2016, the 30-day readmission rate was 11.5% overall. Patients who were readmitted were older with higher incidences of cardiac comorbidities compared with non-readmitted patients. Signiﬁcant risk factors for readmission from the ﬁnal model were the prolonged length of stay, isolated valve surgery, in-hospital complications of sepsis, acute myocardial infarction, diabetes mellitus, gastrointestinal problems wound infection, postoperative acute renal failure, atrial ﬁbrillation (AF), chronic lung disease, obesity, hematocrit <35% before surgery, cardiopulmonary bypass, especially bypass durations of more than 100 minutes.

Perioperative nurses may positively affect reducing readmission rates at different stages of the perioperative continuum of care. All nursing interventions play an important role in minimizing patient risk and preventing or reducing the number of readmissions. Nursing strategies to reduce postoperative cardiac surgery readmission include central line and urinary catheter insertion, cardiopulmonary bypass circuit maintenance, temperature regulation, hair removal, and skin preparation, glycemic control, care of the incision site, treatment and prevention of dysrhythmia, pleural effusion and retained blood syndrome, appropriate discharge teaching, following up with the patients after discharge through telephone conversations and post-discharge care.

Reducing readmission after cardiac surgery remains a quality improvement priority. most readmission risk models examine only coronary artery bypass grafting (CABG). So, this study will be carried out to identify predictors of patients' postoperative readmission after cardiac surgery, including CABG & valvular surgeries.

ELIGIBILITY:
Inclusion Criteria:

* The study will include a sample of 121 adult patients (male and female) who are undergoing CABG or Cardiac Valvular surgeries and whose age is from 18 to 65 years old.

Exclusion Criteria:

* Failed surgery
* Psychiatric patient
* Patient refusal to participate in the study
* Aortic surgeries

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include a sample of 121 adult patients (male and female) who are undergoing CABG or Cardiac Valvular surgeries and whose age is from 18 to 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
detect perioperative risk factors for hospital readmission in patients whose undergoing cardiac surgeries | baseline
  analysis of pre, intra and postoperative risk factors that may cause readmission for patients undergoing Valvular surgery or Coronary artery bypass grafting (CABG)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ali Almasry, Ass.Prof, Study Director — Assistant professor of medical surgical nursing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iribarne A, Chang H, Alexander JH, Gillinov AM, Moquete E, Puskas JD, Bagiella E, Acker MA, Mayer ML, Ferguson TB, Burks S, Perrault LP, Welsh S, Johnston KC, Murphy M, DeRose JJ, Neill A, Dobrev E, Baio KT, Taddei-Peters W, Moskowitz AJ, O'Gara PT. Readmissions after cardiac surgery: experience of the National Institutes of Health/Canadian Institutes of Health research cardiothoracic surgical trials network. Ann Thorac Surg. 2014 Oct;98(4):1274-80. doi: 10.1016/j.athoracsur.2014.06.059. Epub 2014 Aug 28. PMID 25173721
- [Background] Seifert PC. Reducing Readmissions After Coronary Artery Bypass Grafting. AORN J. 2017 Oct;106(4):332-337. doi: 10.1016/j.aorn.2017.08.009. No abstract available. PMID 28958319
- [Background] Ferraris VA, Ferraris SP, Harmon RC, Evans BD. Risk factors for early hospital readmission after cardiac operations. J Thorac Cardiovasc Surg. 2001 Aug;122(2):278-86. doi: 10.1067/mtc.2001.114776. PMID 11479500
- [Background] Demissie, D. B., Doge, G., & Werba, T. B. (2023). The Magnitude of 30-Day Readmission and Factors Associated with Patients Underwent Cardiac Surgery in Tikur Anbessa Specialized Hospital Cardiac Center, Ethiopia. Research Reports in Clinical Cardiology, Volume 14, 35-48. https://doi.org/10.2147/rrcc.s407183
- [Background] Stephens RS, Whitman GJ. Postoperative Critical Care of the Adult Cardiac Surgical Patient. Part I: Routine Postoperative Care. Crit Care Med. 2015 Jul;43(7):1477-97. doi: 10.1097/CCM.0000000000001059. PMID 25962078